CLINICAL TRIAL: NCT05515952
Title: Interleaved TMS-fMRI for Hippocampal Stimulation: Modeling Dose-Response Relationship in Amnestic Mild Cognitive Impairment
Acronym: TMS-fMRI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Ying-hui Chou, Principle Investigator, University of Arizona
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: R21AG077153 (NIH); R21AG077153 (NIH)
Record Dates: First submitted 2022-08-16; First posted 2022-08-25 (Actual); Results first posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Mild Cognitive Impairment
Keywords: Mild Cognitive Impairment; Transcranial Magnetic Stimulation
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Active TBS-Sham TBS (Other): Active TBS in block one, Sham TBS in block two
  Interventions: Device: Transcranial Magnetic Stimulation; Device: Transcranial Magnetic Stimulation (Sham)
- Sham TBS-Active TBS (Other): Sham TBS in block one, Active TBS in block two
  Interventions: Device: Transcranial Magnetic Stimulation; Device: Transcranial Magnetic Stimulation (Sham)

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation — TMS is a non-invasive brain stimulation technique. The primary aim of the study will be to verify the deliverability of the TMS effect on the hippocampus and determine which stimulation protocol is more beneficial to each participant.
Device: Transcranial Magnetic Stimulation (Sham) — TMS is a non-invasive brain stimulation technique. The primary aim of the study will be to verify the deliverability of the TMS effect on the hippocampus and determine which stimulation protocol is more beneficial to each participant. For sham, the side of the coil that does not deliver pulses will be used.

SUMMARY:
Emerging evidence indicates that dysfunction of hippocampal synaptic plasticity, which precedes neuronal degeneration during the progression of Alzheimer's disease (AD), underlies the hallmark cognitive impairment. Although there are currently no effective disease modifying treatments for AD, recent preclinical studies in animal models of AD have suggested that repetitive transcranial magnetic stimulation (rTMS) promotes hippocampal synaptic plasticity and, ultimately, improves learning and memory abilities. Interleaved TBS-MRI is a paradigm, which allows the investigators to study human brain functionality with real-time MRI, to better understand modulations of brain activity in response to the non-invasive brain stimulation, TBS. The interleaved TBSfMRI paradigm can more accurately estimated the immediate brain activity compared to the offline TBS-MRI studies in which TBS is applied outside the MRI. With this interleaved TBS-MRI approach, the investigators will be able to measure immediate changes in targeted brain activity, such as hippocampus activation, following each TBS session. This approach has created the unprecedented potential enabling the investigators to model the dose-dependent effects of TBS more accurately on brain function.

DETAILED DESCRIPTION:
The overarching goal of this proposed project is to maximize TBS effects to non-invasive spaced TBS in MCI. For the comparison, the investigators will include cognitively normal adults. There will be a screening session plus three consecutive days including baseline outcome measures on Day 1, TMS interventions and outcome measures on Day 2, and follow-up measurements on Day 3. In this project, on Day 2, participants will receive three TBS blocks inside the MRI scanner with each TBS block separated by 30-90 minutes to enhance the possibility of maximizing the TBS effect. This will be repeated in two blocks, each with a different TMS protocol. The protocols will be in randomized order.

ELIGIBILITY:
Inclusion Criteria:

* Age 50-80 years
* MCI clinical criteria: (a) self- or informant-reported cognitive complaint; (b) preserved independence in functional abilities; and (c) absence of dementia.
* Objective cognitive impairment supported by the following measures of general cognitive function: (a) Mini-Mental State Exam (MMSE) 24-27 (inclusive); (b) Montreal Cognitive Assessment (MoCA) 18-26 (inclusive); or (c) Clinical Dementia Rating Scale score of 0.5.
* Right handed
* English speaking
* Able to attend daily intervention (Monday-Friday) for 4 days
* Not enrolled in another interventional study within 6 months prior to beginning this study

Exclusion Criteria:

* Contraindications to transcranial magnetic stimulation (TMS) or magnetic resonance imaging (MRI)
* Other neurological disorders (e.g. stroke, head injuries, or multiple sclerosis)
* Untreated depression
* Current cancer treatment or other medical problems that might independently affect cognitive function
* Clinical Dementia Rating Scale score more than 1.0

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ying-hui Chou, ScD, Principal Investigator — University of Arizona
Locations (1):
- Bioscience Research Laboratory, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Active TBS-Sham TBS: Participants first received active stimulation in block 1 and sham in block 2
  Transcranial Magnetic Stimulation: TMS is a non-invasive brain stimulation technique. The primary aim of the study will be to verify the deliverability of the TMS effect on the hippocampus and determine which stimulation protocol is more beneficial to each participant.
  Transcranial Magnetic Stimulation (Sham): TMS is a non-invasive brain stimulation technique. The primary aim of the study will be to verify the deliverability of the TMS effect on the hippocampus and determine which stimulation protocol is more beneficial to each participant. For sham, the side of the coil that does not deliver pulses will be used.
- Sham TBS-Active TBS: Participants received Sham TBS in block 1 and Active in block 2.
  Transcranial Magnetic Stimulation: TMS is a non-invasive brain stimulation technique. The primary aim of the study will be to verify the deliverability of the TMS effect on the hippocampus and determine which stimulation protocol is more beneficial to each participant.
  Transcranial Magnetic Stimulation (Sham): TMS is a non-invasive brain stimulation technique. The primary aim of the study will be to verify the deliverability of the TMS effect on the hippocampus and determine which stimulation protocol is more beneficial to each participant. For sham, the side of the coil that does not deliver pulses will be used.
Period: Block 1
Arm/Group | Active TBS-Sham TBS | Sham TBS-Active TBS
Started | 13 | 12
Completed | 13 | 11
Not Completed | 0 | 1
Period: Washout (1 Month)
Arm/Group | Active TBS-Sham TBS | Sham TBS-Active TBS
Started | 13 | 11
Completed | 11 | 9
Not Completed | 2 | 2
Period: Block 2
Arm/Group | Active TBS-Sham TBS | Sham TBS-Active TBS
Started | 11 | 9
Completed | 11 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active TBS-Sham TBS | Sham TBS-Active TBS | Total
Number analyzed (Participants) | 11 | 9 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 3 | 8
  >=65 years | 6 | 6 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.82 (8.73) | 66.42 (4.64) | 67.19 (7.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 4 | 13
  Male | 2 | 5 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 11 | 8 | 19
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 11 | 9 | 20
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 11 | 9 | 20

OUTCOME MEASURES:

1. Primary Outcome: Correction Rate in Memory Association Recall
Description: Memory tasks will be implemented and measure the correct rate to assess memory function. The scale is the Face Name Associated Memory Score, and the min/max values are 0-1. A higher score indicates a better outcome.
Time Frame: Immediately after intervention day (block 1 day 2) and (block 2 day 2) vs. Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Active TBS: Transcranial Magnetic Stimulation: TMS is a non-invasive brain stimulation technique. The primary aim of the study will be to verify the deliverability of the TMS effect on the hippocampus and determine which stimulation protocol is more beneficial to each participant.
- Sham TBS: Transcranial Magnetic Stimulation (Sham): TMS is a non-invasive brain stimulation technique. The primary aim of the study will be to verify the deliverability of the TMS effect on the hippocampus and determine which stimulation protocol is more beneficial to each participant. For sham, the side of the coil that does not deliver pulses will be used.
Arm/Group | Active TBS | Sham TBS
Number analyzed (Participants) | 20 | 20
units on a scale | .106 (.097) | .031 (.083)

ADVERSE EVENTS:
Time Frame: ~1 year, 5 months
Arm/Group | Active TBS | Sham TBS
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 0/22 | 1/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active TBS (N=22) | Sham TBS (N=22)
Scalp tingling/pressure (Nervous system disorders) | 0 (0) | 1 (1) — Brief (under 1hr) sensation of scalp tingling/pressure at stimulation site with no lingering effects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-03-25): https://cdn.clinicaltrials.gov/large-docs/52/NCT05515952/Prot_SAP_000.pdf